CLINICAL TRIAL: NCT01777087
Title: Brain Imaging of Pain Phenotype and Genotype With Novel Scanning Techniques
Brief Title: Functional Brain Imaging of Pain Phenotype and Genotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jim Ibinson, MD, PhD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO12050474
Record Dates: First submitted 2013-01-10; First posted 2013-01-28 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Pain; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Pain | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy normal volunteers (Experimental): Healthy normal volunteers
  Interventions: Other: gauze soaked with capsaicin

INTERVENTIONS:
Other: gauze soaked with capsaicin — This is a basic science study determining the brain activation that results from painful stimulation. All subjects will have the same painful stimulations and brain images collected.

SUMMARY:
This study has two purposes: first, to locate and identify the "brain activation" (the areas of the brain) which respond to pain; and second, to look at how brain activation is influenced by a person's genetics (the traits they inherited from their parents). A Magnetic Resonance Imaging (MRI) scanner will be used to gather pictures of the brain (similar to an x-ray, but based on different scientific principles) that will be used to determine which areas are active. The hypothesis is that the variation in brain activity between people can be partially explained by genetic differences. This study consists of an two pain tasks applied during a one time visit to the MRI suite. There are no followup visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50
* Right-handed
* Male or female
* Healthy individuals not taking any medication.

Exclusion Criteria:

* Pregnancy
* Diagnosed with any treated or untreated medical or neurological conditions
* Using any prescription drugs, including antidepressants, pain medications, sedative medications, blood pressure medications, seizure medications, or antipsychotics. Oral contraceptives are permitted
* Using any over-the-counter medications including aspirin, Tylenol, or herbal supplements
* Using any illicit substances
* Contraindications to magnetic resonance imaging.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Areas of brain activity from a transcutaneous painful stimulation | At the conclusion of the 1 hour scanning session; Visit one
  A nerve stimulator will be turned on at the level that causes you to report 7/10 pain for 30 seconds, followed by a 30 second period of rest. This will be repeated four times. The areas of brain activity are determined at the end of the 1 hour scanning session by analyzing the brain images. There are no additional followup or long term outcomes.
Areas of brain activity from a 45 minutes Capsaicin cream application | At the conclusion of the 1 hour scanning session; Visit 1
  The painful stimulation will now be caused by placing a piece of gauze soaked with capsaicin, the active ingredients in chili peppers, on the subject's right arm. The areas of brain activity are determined at the end of the 1 hour scanning session by analyzing the brain images. There are no additional followup or long term outcomes.

SECONDARY OUTCOMES:
Pain phenotyping | After the 45 minute Capsaicin cream application; Visit 1
  Subjects will report their pain at least every 3 minutes during the cream application. The subject's pain phenotype will be determined from this response.

CONTACTS AND LOCATIONS:
Overall Officials: James W Ibinson, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Balaban CD, McBurney DH, Affeltranger MA. Three distinct categories of time course of pain produced by oral capsaicin. J Pain. 2005 May;6(5):315-22. doi: 10.1016/j.jpain.2005.01.346. PMID 15890633
- [Background] Campbell CM, Edwards RR, Carmona C, Uhart M, Wand G, Carteret A, Kim YK, Frost J, Campbell JN. Polymorphisms in the GTP cyclohydrolase gene (GCH1) are associated with ratings of capsaicin pain. Pain. 2009 Jan;141(1-2):114-8. doi: 10.1016/j.pain.2008.10.023. Epub 2008 Dec 9. PMID 19081190